CLINICAL TRIAL: NCT05658952
Title: Angio- or Microcatheter- Quantified FFR Virtual PCI Versus Angio-guided PCI in the Achievement of an Optimal Post-PCI FFR
Brief Title: Physiology Optimized Versus Angio-guided PCI
Acronym: AQVA-II
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital of Ferrara (Other)
Responsible Party: Principal Investigator, Gianluca Campo, Study Chair, University Hospital of Ferrara
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 828/2022/DispAOUFe
Record Dates: First submitted 2022-12-01; First posted 2022-12-21 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-12

CONDITIONS: Coronary Artery Disease; Percutaneous Coronary Intervention
Keywords: Percutaneous coronary intervention; Fractional Flow Reserve; Virtual PCI plan
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Intervention Model Description: two nested, randomized, multicenter, open-label trials
Who Masked: Outcomes Assessor
Masking Description: The Independent Clinical Event Committee will perform the blinded adjudication of the events. The Independent Angiography and Physiology Core-lab will perform the primary endpoint analysis
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Angiography-guided PCI (Active Comparator): Patients will receive PCI according to the interpretation of angiography findings by the Interventional Cardiologist.
  Interventions: Other: Angiography-guided PCI
- Microcatheter-derived FFR (Experimental): Patients will receive PCI according to the plan derived from the interpretation of the FFR pullback obtained with microcatheter FFR performed by the Interventional Cardiologist before and after PCI.
  Interventions: Other: Microcatheter-derived FFR
- Angiography-derived FFR (Experimental): Patients will receive PCI according to the plan derived from the interpretation of the FFR pullback obtained with angiography-derived FFR performed by the Interventional Cardiologist before PCI. The angiography-derived FFR can be repeated after PCI to check the results and eventually apply correcting maneuvers.
  Interventions: Other: Angiography-derived FFR

INTERVENTIONS:
Other: Microcatheter-derived FFR — FFR pullback trace is obtained through the manual retrieval performed after the positioning of the microcatheter FFR in the distal portion of the vessel. The pullback speed should be steady and the overall duration would be between 20 and 40 seconds. Then, the Interventional Cardiologist has to decide the procedural plan according to the pullback trace aiming to obtain an optimal post-PCI result in terms of physiology. FFR with pullback can be repeated after stenting to check and correct the result if needed.
  Arms: Microcatheter-derived FFR
Other: Angiography-derived FFR — FFR pullback trace is automatically obtained after the 3-Dimensional reconstruction of the vessel through angiography derived FFR. Then, Interventional Cardiologist has to decide the procedural plan according to the pullback result aiming to obtain an optimal post-PCI result in terms of physiology. Angiography-derived FFR can be repeated after stenting to check and correct the result if needed.
  Arms: Angiography-derived FFR
Other: Angiography-guided PCI — Interventional Cardiologist will perform PCI plan according to his/her the evaluation of angiography.
  Arms: Angiography-guided PCI

SUMMARY:
Angiography-derived Fractional Flow Reserve (FFR) Virtual Percutaneous Coronary Intervention (PCI) plan is superior to conventional angiography-guided PCI in obtaining a good final physiology result, which is, in turn, associated with better prognosis. This has been demonstrated in a population with a relatively low lesion complexity.

Therefore, whether angiography-based FFR virtual PCI could guarantee the same results in some complex anatomical settings (tortuous or calcific vessels, tandem or bifurcation lesions) is not known, also given the inherent limitations of the 3Dimensional (3D)-reconstruction.

The ability of invasive FFR to achieve the same result if compared to angiography-guided PCI has been questioned by recent studies. Recent technological developments, namely the design of pressure wire microcatheters may allow an easier handling of the procedural planning and guidance.

The rationale of the AQVA II study is to test whether a longitudinal FFR-based virtual PCI either angio- or microcatheter- derived is able to improve the post-PCI physiology value if compared to angio-guided PCI in complex and high-risk indicated procedures (CHIP).

DETAILED DESCRIPTION:
Despite the accumulating evidence regarding functional indices utility in setting the indication to and planning percutaneous coronary interventions (PCI), the use of functional assessment in clinical practice is still limited. This is especially true in the post-PCI setting, probably due to lack of evidence and/or specific guidelines/recommendations on how to "react" to a suboptimal post-PCI functional result.

New indices and tools have been developed in an effort to overcome the barriers to a widespread adoption of functional assessment.

All these technological advances brought physiology to a new level transitioning from a binary interpretation of the functional evaluation - positive or negative - to a longitudinal analysis of the whole vessel. The reconstruction of a "physiological map" enables to quantify the physiological impact of each coronary segment/lesion and to identify the mechanisms underlying the suboptimal physiology result at the vessel level. This ability can be translated in simple manoeuvres able to improve the final physiology results and then the patient's prognosis.

The inherent limit of post-PCI physiology is to add measurement and consequent actions after the end of the procedure and not upfront. In addition, it is associated with the increase in procedural time and costs. Thus, a broad application of post-PCI physiology, although clinically meaningful, is difficult.

On the contrary, the systematic application of angiography-derived FFR before stenting to simulate PCI results according to different treatment strategies (virtual PCI) would be an interesting alternative to achieve a fully physiology-guided and optimized procedure. The powerful technological development lays in the possibility to simulate the treatment of one or more lesion, in order to estimate the residual functional value post-PCI: the so-called virtual PCI. These tools are particularly effective in multi-vessel disease patients and in tandem serial stenosis, allowing to individualize the treatment of those lesions related to poor clinical outcomes and avoiding superfluous coronary interventions.

The advantages of a virtual PCI strategy based on angiography-derived FFR application are:

* simple tool, based on what the operator already performs before PCI (namely one or two perpendicular angiographic projections) and not requiring wire or adenosine;
* enables to obtain a longitudinal physiologic map of the vessel with a point-by-point detailed information of the individual impact of any given stenosis;
* simulate the treatment of one or more lesions (virtual PCI) in order to estimate the final functional value post-PCI.

The "Angio-based Quantitative flow ratio (QFR) Virtual PCI versus Conventional Angio-guided PCI in the achievement of an optimal post-PCI QFR" (AQVA)-I trial was the first step toward this direction. The AQVA was a multicenter, investigator-driven, randomized, controlled, parallel group clinical trial. Patients with evidence of angiographically critical coronary lesions and indication to PCI were randomized 1:1 to either angiography-derived FFR virtual PCI or conventional angiography-based PCI. The study aimed to demonstrate the superiority of the angiography-derived FFR virtual PCI over the angiography-based PCI at obtaining an optimal post-PCI result (as defined as a post-PCI QFR value ≥0.90).

From February to December 2021, 300 patients met all inclusion and exclusion criteria and were randomized, for a total of 356 study vessels.

Overall, 38 (10.7%) vessels missed the prespecified post-PCI angiography-derived FFR target (≥0.90). The primary outcome occurred significantly more frequently in the angio-based PCI group (n=26, 15.1%) when compared with the virtual PCI group (n=12, 6.6%; absolute difference 8.5%, relative difference 57%, confidence interval 2.2% - 15.0%, p=0.009). The Δ between pre- and post-PCI physiology value was higher in the virtual PCI groups if compared to the angiography-based group with borderline statistical significance (0.29 [0.23-0.37] versus 0.27 [0.20-0.36], p=0.05).

There were no significant differences among procedural secondary endpoints, such as procedural duration, contrast dye and x-ray utilization. Stent length/lesion and stent number/patient were numerically lower in the virtual PCI group (1 [1-2]; 1.4±0.6 vs 1 [1-2] 1.6±0.7, p=0.06 and 40 [25-55]; 42.7±20.1 vs 44 [28-60]; 46.1±23.1, p=0.08, respectively) whereas procedure length was numerically higher in the virtual PCI group (66 [51-82]; 69±23.1 vs 67 [57-88]; 73.9±23.9, p=0.06). Therefore, virtual PCI based on angiography-derived FFR represents the actual standard of care to guarantee an optimal result in terms of physiology.

The present AQVA-II trial represents the next step of the same approach towards more complex lesions settings.

Patients with severe coronary artery disease at high procedural risk because of comorbidities, complexity of coronary anatomy, and/or poor hemodynamic represent an understudied and underserved patient population.

One of the main limitations of the AQVA-I trial is the absence of a strict inclusion criteria regarding complex and high risk indicated procedures (CHIP)-like lesions (5). The only suggestion was to include long lesions (> 20 mm). Even though, 64 (18%) of included lesions were < 20 mm partially diluting the advantage of the tested strategy. This is confirmed by the high median post-PCI QFR value in both groups (0.97 [0.94-1]). In the study group, namely patients undergoing virtual PCI, the degree of lesions complexity was overall low. The relative simplicity of the lesions included in the AQVA-I trial raises doubts about the validity of the results in contexts of greater complexity, where optimal PCI planning and tools might be different.

Different rapid exchange microcatheters have been developed for FFR assessment. Microcatheters have an ultra-thin profile and they have been designed to allow a rapid exchange system on work-horse wire and easy handling of complex lesions.

As compared to wire-based FFR systems, the potential main advantages of microcatheter-based FFR are:

* Advancement over any traditional 0.014" coronary guidewire;
* The position of the work-horse wire can be maintained during all the procedure, even during pullbacks and post-PCI assessment;
* Tortuous vessels, ostial and/or challenging lesions can be crossed with the work-horse wire and investigated without the need of additional wiring;
* No need for disconnection and reconnection of cable during procedures;
* Less occurrence of clinically significant drift (due to the incorporation of an optical pressure sensor).

To sum up, FFR microcatheter enables to carry out functional evaluations in complex anatomies scenarios (tortuous or calcific vessels, tandem or bifurcation lesions).

At the moment, while microcatheter FFR can be a game changer in vessels with tortuosity, in long challenging diseases, in ostial lesions, and in patients with several comorbidities, there is no clear evidence in this regard. In the same way, no evidence supports the reliability of microcatheter FFR in the post-PCI assessment. Another current current gap in knowledge is to demonstrate that the technical superiority, as compared to wire-based systems, permits to apply a full physiology guided PCI in all anatomical and clinical subsets.

Furthermore, a potential disadvantage is that the microcatheter may increase the degree of coronary artery stenosis and affects the measured FFR value. The influence of the microcatheter on coronary hemodynamic may also be lesion dependent and the small amount of available data might not be translated across a spectrum of vessel and lesion types. A large, dedicated, randomized trial is needed to overcome these issues.

Solid data coming from large randomized controlled trials about microcatheter technology are missing in literature. To date, three studies have been published comparing FFR measured with pressure microcatheter to FFR measured with a pressure wire.

The AQVA-II trial is a program of two nested, randomized, multicenter, open-label trials in Italy. AQVA-II strategy compares longitudinal FFR- versus conventional angiography guided PCI. AQVA-II physiology compares microcatheter- versus angiography-derived FFR guidance.

The primary outcome for AQVA-II strategy is post-PCI FFR >0.86 (superiority). The primary outcome for the AQVA-II physiology is the post-PCI FFR value (non-inferiority).

The Sponsor of the study is U.O. Cardiologia, Azienda Ospedaliero Universitaria di Ferrara. Coordinating center will be the Ferrara University Hospital.

Institutional review board will be obtained in all participating centers. The AQVA trial will be performed in Ferrara University Hospital, Ferrara, Italy. Any additional site participating in the trial will be reported on the website in the dedicated area. The Executive Committee of the Study is composed by Simone Biscaglia (Principal Investigator), Gianluca Campo (Study Chair), Carlo Penzo, Carlo Tumscitz, Andrea Erriquez. The statistical analysis will be performed by the Centre for Epidemiology and Statistics of the University of Ferrara (Elisa Maietti, Stefano Volpato).

ELIGIBILITY:
Inclusion Criteria:

1. Indication to PCI for either acute or chronic coronary syndrome
2. Signed informed consent
3. At least one of the following CHIP lesion characteristic:

   * Long lesion (>28 mm);
   * Tandem lesions;
   * Severe calcifications;
   * Severe tortuosity;
   * True bifurcation lesions: involving a significant (> 50%) diameter stenosis both in the main vessel and side branch (i.e. MEDINA 1,1,1; 1,0,1; or 0,1,1) and with a relevant side branch, namely ≥2.00 mm;
   * In-stent restenosis (ISR).
   * Left main stem disease.

Exclusion Criteria:

1. Planned surgical revascularization
2. Prior Coronary Artery Bypass Graft (CABG) Surgery
3. Culprit lesion of STEMI or NSTEMI
4. Revascularization of a chronic total occlusion
5. Non-cardiovascular co-morbidity reducing life expectancy to < 1 year
6. Any factor precluding 1-year follow-up

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 305 (Actual)
Dates: Start 2022-12-01 (Actual); Primary Completion 2023-06-20 (Actual); Study Completion 2024-12-07 (Actual)

PRIMARY OUTCOMES:
Post-PCI Fractional Flow Reserve (FFR) | at the end of the procedure (at the moment of the last angiography)
  At the end of the procedure in all patient a blinded invasive post-PCI FFR will be obtained

SECONDARY OUTCOMES:
VOCE | 1 year
  vessel-oriented composite endpoint (VOCE), defined as the composite of vessel-related cardiovascular death, vessel-related myocardial infarction (MI), and ischemia-driven target vessel revascularization (TVR).
Post-PCI Distal Pressure (Pd) / Aortic Pressure (Pa) | at the end of the procedure (at the moment of the last angiography)
  At the end of the procedure in all patient a blinded invasive post-PCI Pd/Pa will be obtained

CONTACTS AND LOCATIONS:
Locations (2):
- Italy (2):
  - University Hospital of Ferrara, Cona, Ferrara
  - Santa Maria Goretti Hospital, Latina, LT

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Biscaglia S, Verardi FM, Erriquez A, Colaiori I, Cocco M, Cantone A, Pompei G, Marrone A, Caglioni S, Tumscitz C, Penzo C, Manfrini M, Leone AM, Versaci F, Campo G. Coronary Physiology Guidance vs Conventional Angiography for Optimization of Percutaneous Coronary Intervention: The AQVA-II Trial. JACC Cardiovasc Interv. 2024 Jan 22;17(2):277-287. doi: 10.1016/j.jcin.2023.10.032. Epub 2023 Oct 23. PMID 37902150
- [Derived] Marrone A, Erriquez A, Verardi FM, Colaiori I, Cocco M, Caglioni S, Tumscitz C, Penzo C, Marchini F, Meinen J, McNutt J, Buijs JOD, Chiu WC, Versaci F, Campo G, Biscaglia S. Additional Value of Optical Coherence Tomography-Derived Virtual Flow Reserve for Percutaneous Coronary Intervention Guidance. Catheter Cardiovasc Interv. 2025 Dec;106(7):3456-3464. doi: 10.1002/ccd.70207. Epub 2025 Sep 23. PMID 40988408